CLINICAL TRIAL: NCT05821179
Title: Salivary LINC00657 as a Diagnostic Biomarker for Oral Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Nayroz Tarrad, associate professor, Fayoum University
Other Study IDs: M1
Record Dates: First submitted 2023-03-26; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Oral squamous cell carcinoma, oral potentially malignant disorders, saliva, LINC00657, miR-106a.
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: 12 patients diagnosed with OSCC.
- Group II: 12 patients diagnosed with OLP.
- Group III: 12 systemically free individuals with no oral mucosal lesions.

SUMMARY:
This study was designed to verify the role of salivary LINC00657 as a diagnostic marker in oral squamous cell carcinoma (OSCC) patients as compared to oral lichen planus (OLP) (as an example of oral potentially malignant lesions) and normal individuals, and to show its relation to miR-106a. A total of 36 participants were included.

DETAILED DESCRIPTION:
This study was designed to verify the role of salivary LINC00657 as a diagnostic marker in oral squamous cell carcinoma (OSCC) patients as compared to oral lichen planus (OLP) (as an example of oral potentially malignant lesions) and normal individuals, and to show its relation to miR-106a. A total of 36 participants were included, subdivided into 3 groups: Group I: 12 patients diagnosed with OSCC. Group II: 12 patients diagnosed with OLP. Group III: 12 systemically free individuals with no oral mucosal lesions. statistical analysis and ROC analysis were performed

ELIGIBILITY:
Inclusion Criteria:

* group I : oral squamous cell carcinoma lesions (OSCC)
* group II: oral lichen planus lesions (OLP)
* group III: systemically healthy volunteers

Exclusion Criteria:

* oral lesions other than OSCC / OLP in group I and II
* any oral lesion in group III
* pregnant females

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - patients recruited from the outpatient clinic of departments of oral diagnosis and medicine and periodontology Fayoum, Beni-Suef and Ahram-Candian universities
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
LINC00657 level in salivary samples from all participants measured using PCR | level of miR-106a is measured after the completion of all salivary sample collection carried at the 1 day of enrollment of subjects in the investigation after diagnosis confirmation
  quantitative real-time PCR is used to detect LINC00657 levels in saliva samples from patients with OSCC and OPMD compared to healthy subjects

SECONDARY OUTCOMES:
miR-106a level in salivary samples from the included subjects evaluated by PCR | level of miR-106a is measured after the completion of all salivary sample collection carried at the 1 day of enrollment of subjects in the investigation
  quantitative real-time PCR is used to detect miR106a levels in saliva samples from patients with OSCC and OPMD compared to healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Nayroz Tarrad, as. professor, Principal Investigator — faculty of dentistry, Fayoum university
Locations (1):
- faculty of dentistry, Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tarrad NAF, Hassan S, Shaker OG, AbdelKawy M. "Salivary LINC00657 and miRNA-106a as diagnostic biomarkers for oral squamous cell carcinoma, an observational diagnostic study". BMC Oral Health. 2023 Dec 12;23(1):994. doi: 10.1186/s12903-023-03726-0. PMID 38087258